CLINICAL TRIAL: NCT01333566
Title: Qigong Exercise May Benefit Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11889
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental)
  Interventions: Behavioral: Intervention Group
- Control Group (Placebo Comparator)
  Interventions: Behavioral: Placebo Comparator: Control Group

INTERVENTIONS:
Behavioral: Intervention Group — The study will include one week baseline phase, 6-week intervention phase, and a 3-month follow-up evaluation. Subjects in the intervention group will go through three training sessions during the baseline phase, weekly group exercise sessions once per week and daily home exercises two times each day during the intervention phase, and a follow-up evaluation in three months after the intervention phase.
  Arms: Intervention Group
Behavioral: Placebo Comparator: Control Group — Subjects in the control group will be monitored during the baseline and intervention phase without participating in the interventional exercise. At the end of intervention phase, the subjects will have the option to stop their participation or switch to the intervention group.
  Arms: Control Group

SUMMARY:
The long-term goal of our research program is to develop an effective and cost-saving mind-body therapy to help patients with FM. The objective of this pilot study is to gather pilot data of the effect on pain, fatigue, sleep quality, and quality of life in FM patients using a specific type of qigong exercise, i.e. "six healing sound" qigong. Changes in relevant brain activity will be monitored in study subjects before and after the qigong exercise program, which may help us in better understanding the underlying mechanism of the qigong exercise. Data collected in this pilot study will help the investigators in preparation for a future clinical trial with a larger sample size. Our central hypothesis for the future clinical trial is that qigong exercise will lead to a significantly greater improvement in pain, fatigue, sleep quality, and quality of life in the experimental group compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of primary FM, based on the 1990 American College of Rheumatology criteria (Wolfe et al, 1990),
* between the ages of 18 and 70 years;
* willing to withdraw from CNS-active therapies commonly used to treat FM; willing to discontinue treatment with transcutaneous electrical nerve stimulation, biofeedback, tender- and trigger-point injections, acupuncture, and anesthetic or narcotic patches;
* with a raw score > 4 on the physical function component of the Fibromyalgia Impact Questionnaire (FIQ) (Burckhardt et al, 1991);
* and a mean visual analog scale (VAS) pain score > 40 on a scale from 0 to 100.

Exclusion Criteria:

* severe psychiatric illness;
* a current major depressive episode (as determined by a Beck Depression Inventory (Beck et al, 1961) score >25);
* significant suicide risk;
* abuse of alcohol, benzodiazepines, or other drugs; a history of behavior that would prohibit compliance for the duration of the study;
* active cardiovascular, pulmonary, hepatic, renal, gastrointestinal, or autoimmune disease (except Hashimoto's or Graves' disease that had been stable for 3 months before screening);
* current systemic infection; active cancer (except basal cell carcinoma); unstable endocrine disease; severe sleep apnea;
* prostate enlargement or other genitourinary disorder (male patients);
* or pregnancy or breastfeeding (female patients).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of qigong exercise on pain | up to 3months

SECONDARY OUTCOMES:
To investigate the effect of qigong exercise on fatigue | up to 3 months
To investigate the effect of qigong exercise on sleep quality | up to 3 months
To investigate the effect of qigong exercise the quality of life in FM patients. | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wen Liu, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University Of Kansas Medical Center, Kansas City, Kansas, United States